CLINICAL TRIAL: NCT03847532
Title: Diagnosis and Treatment of Russian Patients With MutYH-associated Polyposis
Brief Title: MUTYH-associated Polyposis
Acronym: MAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 119
Record Dates: First submitted 2019-01-20; First posted 2019-02-20 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: MutYH-associated Polyposis
Keywords: MutYH-associated polyposis; familial adenomatous polyposis; biallelic mutation; monoallelic mutation; colproctectomy
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Polymerase Chain Reaction; Polymorphism, Single-Stranded Conformational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with mutations in the MutYH-gene (Other): Patients with established diagnosis of MutYH-associated polyposis with monoallelic and biallelic mutations in the MutYH-gene
  Interventions: Genetic: Sanger sequencing method
- Patients with multiple colon polyps (Other): Number of polyps from 4+
  Interventions: Genetic: Sanger sequencing method
- Control sample (Other): Patients who did not have colon polyps
  Interventions: Genetic: Sanger sequencing method

INTERVENTIONS:
Genetic: Sanger sequencing method — Amplification of the examined fragments of the MutYH gene was conducted using the PCR machine TP4-PCR-01-Tertsik (DNA-Technology, Russia) containing 25 μL of the reaction mixture: 0.1-1.0 μg genomic DNA; 0.25 μM of each original oligoprimer; 200 μM of each nucleosidetriphosphate; 1 U Taq polymerase; PCR buffer (500 mM Tris, 500 mM KCl, pH 8.74); 2.5 μL MgCl2 (25 mM)); deionized water; 20-30 μL of mineral oil. For MutYH gene analysis (Transcript ENST00000257430) Primer3 software (http:// frodo.wi.mit.edu/primer3/input.htm) was selected and 16 primer pairs. The variants of the primary structure in the obtained fragments were revealed using SSCP. DNA fragments containing electrophoretically identified variants were sequenced.
  Other Names: polymerase chain reaction; SSCP

SUMMARY:
This is single-center, prospective, non-randomized study

DETAILED DESCRIPTION:
The study will include patients with more than 3 polyps, without mutations in the APC gene. Using molecular genetic research methods (polymerase chain reaction, SSCP, sequencing by Sanger method) mutations in the MutYH gene will be studied. For all patients with mutations in the MutYH gene, an optimal diagnostic algorithm will be developed. The significance of monoallelic mutations in the MutYH gene will be determined. Clinical monitoring will be defined. Optimal amount of surgical intervention will be suggested.

ELIGIBILITY:
Inclusion Criteria:

1. patients with multiple colon polyps (n polyps = 4+)
2. patient consent to participate in the study

Exclusion Criteria:

1. presence of mutations in the APC gene
2. patient's refusal to participate in the study

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-10-10 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Patients with germIine mutations in MutYH | from 0 to 6 months
  number of patients with monoallelic and biallelic mutations in the MutYH-gene

CONTACTS AND LOCATIONS:
Locations (1):
- State Scientific Centre of Coloproctology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No